CLINICAL TRIAL: NCT02030366
Title: A Portable Chromatic Multifocal Pupillometer for Objective Early Detection and Follow-up of Changes in Intracranial Pressure in Patients With Acute Head Injury
Brief Title: Chromatic Multifocal Pupillometer for Detection and Follow-up of Acute Head Injury
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Head of Electrophysiology Service, Sheba Medical Center
Other Study IDs: 9994-12-SMC
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury (TBI) Patients
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI patients
- Healthy Volunteers

SUMMARY:
Traumatic Brain Injury (TBI) is a common injury in combat, terrorist attacks and sports such as football and hockey. Unnecessary delays in the diagnosis and treatment of brain damage in patients who can benefit from evacuation procedures can lead to worse brain injury, worse outcome and, sometimes, unnecessary death. However, there is no reliable and sensitive method for diagnosis of TBI severity in the field. In this study we will examine the feasibility of using this a multifocal chromatic pupillometer for monitoring TBI, by examining the pupillary response to multifocal chromatic stimuli in intracranial pressure (ICP)-monitored severe TBI patients. As control, normal subjects will be tested for pupillary responses using this device.

DETAILED DESCRIPTION:
To examine the feasibility of using the multifocal chromatic pupillometer for monitoring TBI, the pupillary response to multifocal chromatic stimuli will be assessed in 20 healthy subjects and 20 ICP-monitored severe TBI patients.

The portable pupillometer will be tested in 20 healthy volunteers. Their pupillary responses will be measured 3 times/day for 1 week.

Pupillary response of 20 severe TBI patients will be evaluated as detailed below at the following time points:

1. At admittance to ICU, prior to insertion of ICP and CT scan
2. Prior to CT scans that are routinely performed at day 3 and 7 post injury
3. Routinely at the beginning of every medical personnel shift for 7 days (3 times a day).
4. With every change in ICP(more than 5 mmHg for more then 15 min) Data will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects -
* Male or female patients, age between 18 and 70 years, inclusive
* Informed written consent will be obtained from all participants.
* Normal eye examination
* Best-corrected visual acuity (BCVA) of 20/20
* Normal color vision test (Roth-28-hue test)
* Written informed consent to participate in the study,
* TBI-patients:
* Male or female patients, age between 18 and 70 years, inclusive
* Initiation of study before the insertion of the ICP monitor.
* TBI diagnosed by history and clinical examination
* Glasgow Coma Scale (GCS) score between 3 and 8, inclusive
* Evidence of TBI confirmed by abnormalities consistent with trauma on CT scan upon admission (diffuse injury II-IV, evacuated and non-evacuated mass lesion, Marshall's CT Classification)
* Indication for ICP monitoring
* Written informed consent to participate in the study, signed by a family member and independent physician.

Exclusion Criteria:

* Healthy subjects
* History of past or present ocular disease
* Use of any topical or systemic medications that could adversely influence efferent pupil movements
* TBI-patients
* High levels of barbiturate medications as they abolish pupillary responsiveness
* Coma suspected to be primarily due to other causes (e.g. alcohol)
* Preexisting clinically significant disease or chronic condition that can be ascertained at the time of admission and could affect pupillary response or measurement (such as known retinal dystrophy disease, glaucoma or dense cataract.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TBI patients addmitted to Tel Hashomer Intensive Care Unit, and halthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pupillary response at 5 points of Visual field to blue and red light | 7 days
  Pupillary response at 5 points of Visual field to blue and red light will be measured 3 times a day for a week for the health subjects. The TBI patients will be monitored for pupillary response:
  * At admittance to ICU, prior to insertion of ICP and CT scan
  * Prior to CT scans that are routinely performed at day 3 and 7 post injury
  * Routinely at the beginning of every medical personnel shift for 7 days (3 times a day).
  * With every change in ICP(more than 5 mmHg for more then 15 min)

SECONDARY OUTCOMES:
Intra Cranial Pressure | 7 days
  TBI patients only will be continuously monitored for Intra Cranial Pressure (ICP)

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery Department, Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Skaat A, Sher I, Kolker A, Elyasiv S, Rosenfeld E, Mhajna M, Melamed S, Belkin M, Rotenstreich Y. Pupillometer-based objective chromatic perimetry in normal eyes and patients with retinal photoreceptor dystrophies. Invest Ophthalmol Vis Sci. 2013 Apr 17;54(4):2761-70. doi: 10.1167/iovs.12-11127. PMID 23482470